CLINICAL TRIAL: NCT01749215
Title: A Controlled Trial of Topiramate Treatment for Alcohol Dependence in Veterans With PTSD
Acronym: TAP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT110423; W81XWH-11-PHTBI-BAPHA (Other: Department of Defense)
Record Dates: First submitted 2012-11-09; First posted 2012-12-13 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Dependence; Posttraumatic Stress Disorder (PTSD)
Keywords: pharmacotherapy; alcohol dependence; Veterans
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Topiramate; Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Topiramate capsules daily - up to 300 mg
  Interventions: Drug: Topiramate; Behavioral: Medical Management
- Placebo (Placebo Comparator): Placebo capsules daily - up to 300 mg
  Interventions: Drug: placebo; Behavioral: Medical Management

INTERVENTIONS:
Drug: Topiramate — Experimental study drug
  Arms: Topiramate
Drug: placebo — Placebo comparator
  Arms: Placebo
Behavioral: Medical Management — Brief alcohol counseling

SUMMARY:
The goal of this project is to improve the treatment of veterans with co-occurring alcohol dependence and posttraumatic stress disorder (PTSD). The PI and co-investigators will conduct a controlled clinical trial of topiramate for the treatment of these co-occurring disorders.

DETAILED DESCRIPTION:
This project consists of a controlled clinical trial of topiramate treatment to reduce alcohol use and PTSD symptoms in veterans with these co-occurring disorders.

This is a prospective randomized double-blind controlled parallel groups clinical trial of topiramate or or placebo up to 300 mg per day, combined with weekly alcohol counseling, over a 12-week treatment period with a week 16 follow-up. The study population consists of 150 male and female veterans between the ages of 18-69 who have concurrent diagnoses of alcohol use disorder and PTSD. Subjects meet with research staff weekly to receive study medication, manualized alcohol counseling, and research assessments. The primary treatment outcome is the percent of days of drinking; the secondary outcome is PTSD symptom severity. Exploratory measures include assessments of impulsivity and decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female veterans
2. Ages18 to 69 (inclusive)
3. Current DSM-IV diagnosis of PTSD
4. Current (past month) DSM-IV diagnosis of an Alcohol Dependence
5. Level of drinking must meet criteria for "at-risk " or "heavy" drinking by NIAAA threshold (NIAAA 2007): at least 15 standard drinks per week on average over the 4 weeks prior to study entry for men and at least 8 standard drinks per week on average for women.
6. Subjects must express a desire to reduce alcohol consumption with the possible long-term goal of abstinence.
7. Female subjects must have a negative urine pregnancy test and must be either postmenopausal for at least one year, or practicing an effective method of birth control (e.g., surgically sterile, spermicide with barrier, male partner sterilization; or abstinent and agrees to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence)
8. Subjects must have a Breath Alcohol Concentration (BAC) of < 0.02% when signing informed consent.

Exclusion Criteria:

1. Psychotic disorders, bipolar disorder, dementia, or other psychiatric disorders judged to be unstable.
2. Subjects known to have clinically significant unstable medical conditions, including but not limited to:

   * Clinically significant renal disease and/or impaired renal function as defined by clinically significant elevation of blood urea nitrogen (BUN) or creatinine or an estimated creatinine clearance of < 60 mL/min
   * AST and/or ALT >5 times the upper limit of the normal range and/or an increased serum bilirubin >2 times the upper limit of normal.
   * Seizure disorders
3. History of glaucoma.
4. History of kidney stones.
5. Concurrent participation in another treatment study.
6. Female patients who are pregnant or lactating.
7. Current Topiramate use or use within the past 4 weeks.
8. Current medications for alcohol dependence (disulfiram, naltrexone, or acamprosate) or use in the past week.
9. Needing acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD);
10. Subjects who are legally mandated to participate in an alcohol treatment program.
11. Subjects who have had a suicide attempt in the past 6 months or suicidal ideation in the 90 days prior to enrollment.
12. Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate,
13. Subjects with seizure disorders that require anticonvulsant medications
14. Subjects currently being treated with another anticonvulsant.
15. Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the topiramate package insert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 72 | 79
Completed | 47 | 53
Not Completed | 25 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 72 | 79 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 71 | 134
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (12.2) | 52.0 (11.6) | 51.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 62 | 70 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 55 | 65 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 22 | 29 | 51
  White | 33 | 29 | 62
  More than one race | 10 | 12 | 22
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 72 | 79 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Heavy Drinking Days Over the 12 Weeks of Study Treatment as Assessed by the Timeline Followback (TFLB)
Description: Timeline Followback (TLFB) data was recorded using a calendar, with participants providing retrospective reports of daily drinking over the past week(s). The percent of heavy drinking days per week was calculated from the calendar data. The change in percentage of heavy drinking days was calculated by subtracting Week 0 (baseline) data from Week 12. Negative scores indicate improvement.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percent heavy drinking days
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 72 | 79
percent heavy drinking days | -36.2 (0.41) | -25.1 (.36)

2. Secondary Outcome: Change in PTSD Symptom Severity as Assessed by the PTSD Checklist (PCL)
Description: The PCL is a 17-item self-report measure reflecting DSM-IV symptoms of PTSD. A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items that have response options ranging from 1 "Not at all" to 5 "Extremely". It was calculated by subtracting the data collected at Week 0 (baseline) from data collected at Week 12. Negative scores indicate improvement.
Time Frame: Baseline to Week 12
Population: Data were only collected for N=42 for the Topiramate arm and N=49 for the Placebo arm, as reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 42 | 49
score on a scale | -15.4 (14.8) | -15.9 (14.9)

3. Secondary Outcome: Change in Impulsivity as Assessed by Delay Discounting (DD)
Description: DD measures impulsivity by evaluating discount rates for delayed rewards. On a computer screen, the participant is shown hypothetical dollar amounts that could be received immediately, while a hypothetical $100 reward is displayed continuously. The "delay duration" is the waiting period for the $100 delayed reward. The computer randomly presents each immediate reward dollar amount, one at a time and participants are asked to choose between each immediate reward or the delayed $100. The same procedure will be repeated for each of the delay periods. Delay discounting quantifies the devaluation of rewards over time, which allows for an index of overall discounting rate (k). Higher k values indicate greater discounting and therefore greater impulsivity. DD score change was measured by subtracting Week 0 (baseline) scores from Week 12 scores, with negative scores representing improvement.
Time Frame: Baseline to Week 12
Population: Data were only collected for N=22 for the Topiramate arm and N=16 for the Placebo arm, as reported here.
Measure: Mean (Standard Deviation); unit: K-value
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 22 | 16
K-value | -0.020 (0.34) | 0.058 (0.17)

4. Secondary Outcome: Change in Risk-taking Behavior as Assessed by the Balloon Analogue Risk Task (BART)
Description: BART is a computerized measure of risk taking behavior that displays a computer-generated balloon on a computer monitor. Participants gradually pump (inflate) the balloon. Each pump adds 5 cents to a temporary bank. After each pump, participants have 2 options, 1) continue to pump the balloon and risk bursting it, losing all the money from that balloon, or 2) saving the accumulated money to a permanent bank. Whenever a balloon bursts or the participant chooses to bank money, they start with a new balloon. Participants respond to 30 balloons, each having a different bursting point. With each pump, participants weigh the potential gain of collecting more money against the risk of losing all money accumulated with that balloon.
  Greater number of pumps indicates greater risk taking. Change was calculated by subtracting Week 12 scores from Week 0 (baseline), with negative scores representing improvement and positive scores representing worsening risk taking.
Time Frame: Baseline to Week 12
Population: Data were only collected for N=43 for the Topiramate arm and N=46 for the Placebo arm, as reported here.
Measure: Mean (Standard Deviation); unit: Total pumps
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 43 | 46
Total pumps | 26.7 (205.4) | 13.4 (199.0)

5. Secondary Outcome: Change in Decision-making Behavior as Assessed by the Iowa Gambling Task (IGT)
Description: The Iowa Gambling Task (IGT) is a computerized assessment that evaluates decision-making by tracking the selection of advantageous or disadvantageous electronic cards from four decks. Subjects are presented the 4 decks of cards on a computer screen and are told that they can win money by picking cards from the most advantageous deck. After each deck selection, subjects are provided feedback as to whether their selection resulted in a "win" or a "loss" and the dollar amount of the win/loss. Data indicate change from baseline in mean number of cards selected from advantageous decks minus number of cards selected from disadvantageous decks as a function of drug condition. Change measured by substracting Week 0 (baseline) scores from Week 12 scores. Higher numbers indicate better decision making regarding advantageous cards.
Time Frame: Baseline to Week 12
Population: Data were only collected for N=31 for the Topiramate arm and N=34 for the Placebo arm, as reported here.
Measure: Mean (Standard Deviation); unit: test cards
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 31 | 34
test cards | 2.03 (13.80) | 2.80 (14.54)

ADVERSE EVENTS:
Time Frame: Over 16 weeks.
Description: We used the Adverse Event Symptom Checklist at every study visit (Visits 0 - 12 and 16), which assessed the most reported adverse events listed in the FDA Prescribing Information.
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/72 | 1/79
Serious Adverse Events (participants affected / at risk) | 2/72 | 9/79
Other Adverse Events (participants affected / at risk) | 70/72 | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=72) | Placebo (N=79)
Inpatient hospitalization of less than 24 hours with diagnosis of Type 2 MI (Cardiac disorders) | 0 (0) | 1 (1) — This happened in the context of cocaine and methamphetamine use, with discharge within 24 hours.
Inpatient medical hospitalization for alcohol withdrawal. (Nervous system disorders) | 0 (0) | 1 (1)
Inpatient psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported increased suicidal ideation and was willing to voluntarily go to psych emergency services (PES) at the SFVAMC. PES staff conducted their own assessment and concluded inpatient psychiatric hospitalization would be beneficial.
Inpatient psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — The participant voluntarily presented at PES at SFVAMC looking for housing. During routine assessment, participant reported cocaine use, hopelessness and thoughts of self-harm without a specific plan. Determined that needed to be admitted to PICU.
Inpatient medical hospitalization due to abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — The participant was brought by ambulance to the emergency department because of abdominal pain and vomiting. Participant has history of multiple bowel obstructions.
Death of research participant (General disorders) | 0 (0) | 1 (1) — Coroner's report on cause of death: cocaine toxicity
Inpatient hospitalization due to congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1) — Thought to be secondary to hypertension and chronic alcohol use.
Inpatient hospitalization due to suicidal ideation and alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1)
Inpatient hospitalization due to shortness of breath in the setting of abdominal distension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant was experiencing increased shortness of breath in the setting of abdominal distension and 20 pound weight gain over 3 months. Discharge diagnosis was COPD and lactose intolerance.
Inpatient hospitalization for lower quadrant pain, cough and chills (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — It was found that participant had a fever, increased white blood cells, and his lungs were filled with liquid. Veteran was prescribed amoxicillin and clavulonic acid for 7 days to treat aspiration pneumonia.
Inpatient hospitalization for pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inpatient hospitalization for MRSA (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=72) | Placebo (N=79)
Numbness or tingling (Nervous system disorders) | 22 | 13
Change in sense of taste (Nervous system disorders) | 29 | 29
Fatigue (General disorders) | 17 | 17
Loss of appetite (Gastrointestinal disorders) | 38 | 23
Difficulty with concentration or attention (Nervous system disorders) | 7 | 10
Diarrhea (Gastrointestinal disorders) | 30 | 28
Dizziness (Ear and labyrinth disorders) | 17 | 19
Itching (Skin and subcutaneous tissue disorders) | 26 | 21
Sleepiness (General disorders) | 19 | 20
Slow thinking (Nervous system disorders) | 17 | 17
Abnormal vision (Eye disorders) | 23 | 17
Eye pain (Eye disorders) | 16 | 18
Confusion (Nervous system disorders) | 26 | 11
Language problems (e.g., word searching) (Nervous system disorders) | 7 | 13
Depression (Psychiatric disorders) | 9 | 7
Suicidal thoughts or actions (Psychiatric disorders) | 6 | 6
Nervousness (Psychiatric disorders) | 7 | 10
Difficulty with memory (Nervous system disorders) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT01749215/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT01749215/ICF_001.pdf